CLINICAL TRIAL: NCT02026401
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled, Parallel Group, Multiple Center Study to Evaluate the Safety, Tolerability, and Pharmacodynamic Activity of NGM282 in Combination With Ursodeoxycholic Acid (UDCA) Administered for 28 Days in Patients With Primary Biliary Cirrhosis
Brief Title: Phase 2 Study of NGM282 in Patients With Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Collaborators: NGM Biopharmaceuticals Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0103
Record Dates: First submitted 2013-12-30; First posted 2014-01-03 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — aldafermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NGM282 Dose 1 (Experimental): NGM282 Dose 1
  Interventions: Biological: NGM282
- NGM282 Dose 2 (Experimental): NGM282 Dose 2
  Interventions: Biological: NGM282
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NGM282
  Arms: NGM282 Dose 1; NGM282 Dose 2
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and activity of NGM282 in patients with Primary Biliary Cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, between 18 and 75 years of age, inclusive
* PBC diagnosis consistent with AASLD and EASL guidelines
* Stable dose of UDCA

Exclusion Criteria:

* Chronic liver disease of a non-PBC etiology
* Evidence of clinically significant hepatic decompensation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Absolute change in plasma ALP from Baseline to Day 28 | 28 days

SECONDARY OUTCOMES:
Absolute change in bilirubin from Baseline to Day 28 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Rossi, PharmD, Study Director — NGM Biopharmaceuticals, Inc
Locations (17):
- United States (7):
  - NGM Clinical Study Site 103, Phoenix, Arizona
  - NGM Clinical Study Site 108, Coronado, California
  - NGM Clinical Study Site 101, Detroit, Michigan
  - NGM Clinical Study Site 105, Durham, North Carolina
  - NGM Clinical Study Site 102, Dallas, Texas
  - NGM Clinical Study Site 113, San Antonio, Texas
  - NGM Clinical Study Site 104, Richmond, Virginia
- Australia (10):
  - NGM Clinical Study Site 602, Sydney, New South Wales
  - NGM Clinical Study Site 606, Sydney, New South Wales
  - NGM Clinical Study Site 609, Sydney, New South Wales
  - NGM Clinical Study Site 611, Sydney, New South Wales
  - NGM Clinical Study Site 614, Brisbane, Queensland
  - NGM Clinical Study Site 607, Adelaide, South Australia
  - NGM Clinical Study Site 608, Adelaide, South Australia
  - NGM Clinical Study Site 601, Melbourne, Victoria
  - NGM Clinical Study Site 604, Melbourne, Victoria
  - NGM Clinical Study Site 613, Melbourne, Victoria

REFERENCES:
- See also: Related Info — http://www.ngmbio.com